CLINICAL TRIAL: NCT00492453
Title: A Controlled Randomized Trial Comparing Spinal Versus General Anesthesia for Elective Laparoscopic Cholecystectomy in Fit Patients
Brief Title: Spinal Versus General Anesthesia for Laparoscopic Cholecystectomy
Acronym: SALC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Collaborators: Larissa University Hospital (Other)
Responsible Party: George Tzovaras, MD, University of Thessaly, School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UThessaly 9-04
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-06

CONDITIONS: Spinal Anesthesia; General Anesthesia; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Laparoscopic cholecystectomy under spinal anesthesia
  Interventions: Procedure: laparoscopic cholecystectomy
- 2 (Active Comparator): Laparoscopic cholecystectomy under general anesthesia
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — elective laparoscopic cholecystectomy using CO2 pneumoperitoneum under different methods of anesthesia

SUMMARY:
The purpose of the study is to assess whether spinal anesthesia is or not superior to the standard general anesthesia for fit patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy under regional anesthesia alone has been reported only occasionally in the past; all these reports included patients unfit to receive general anesthesia, mainly patients with severe chronic obstructive airway disease. Regional anesthesia has been used for laparoscopy in fit patients almost exclusively in combination with general anesthesia, in order to extend the analgesic effect during the early postoperative period. Surprisingly, in the era of minimally invasive medicine, regional anesthesia has not gained popularity, and has not been routinely used as a sole method of anesthesia in laparoscopic procedures. It is generally accepted that all laparoscopic procedures are merely a change in access and still require general anesthetic; hence the difference from conventional surgery is likely to be small. This statement is predominantly based on the assumption that laparoscopy necessitates endotracheal intubation to prevent aspiration and respiratory embarrassment secondary to the induction of CO2 pneumoperitoneum which in turn is not well tolerated in a patient who is awake during the procedure. However, it is surprising that regional anesthesia has been successfully used for laparoscopic cholecystectomy in patients unfit to have the procedure under general anesthesia, but has not been tested in fit patients, in whom any presumed risk would be, theoretically, much lower. We have recently shown in a pilot study the feasibility to perform successfully and safely laparoscopic cholecystectomy with low pressure CO2 pneumoperitoneum under spinal anesthesia alone, in fit patients with symptomatic gallstone disease. We have also noticed that spinal anesthesia results in exceptionally minimal postoperative pain. After this pilot study, we designed a controlled randomized trial in order to compare spinal anesthesia with the standard general anesthesia for elective laparoscopic cholecystectomy in fit patients.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy
* ASA I, II
* BMI< 30
* normal coagulation profile

Exclusion Criteria:

* acute cholecystitis / cholangitis / pancreatitis
* previous open surgery in the upper abdomen
* contraindication for pneumoperitoneum
* contraindication for spinal anesthesia (ie spinal deformity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 24hrs

SECONDARY OUTCOMES:
complications | 30 days
hospital stay | time from intervention to discharge
patient satisfaction | within 2 weeks from intervention

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Hatzitheofilou, MD, Study Chair — University of Thessaly, School of Medicine; George Tzovaras, MD, Study Director — University of Thessaly, School of Medicine; Frank Fafoulakis, MD, Principal Investigator — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Tzovaras G, Fafoulakis F, Pratsas K, Georgopoulou S, Stamatiou G, Hatzitheofilou C. Laparoscopic cholecystectomy under spinal anesthesia: a pilot study. Surg Endosc. 2006 Apr;20(4):580-2. doi: 10.1007/s00464-005-0405-1. Epub 2006 Jan 25. PMID 16437265
- [Result] Tzovaras G, Fafoulakis F, Pratsas K, Georgopoulou S, Stamatiou G, Hatzitheofilou C. Spinal vs general anesthesia for laparoscopic cholecystectomy: interim analysis of a controlled randomized trial. Arch Surg. 2008 May;143(5):497-501. doi: 10.1001/archsurg.143.5.497. PMID 18490561